CLINICAL TRIAL: NCT07005934
Title: Effects of Percussion Therapy on the Biomechanics of Pickleball Movement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Point Loma Nazarene University (Other)
Collaborators: Therabody, Inc. (Industry)
Responsible Party: Principal Investigator, Arnel Aguinaldo, Full Professor, Point Loma Nazarene University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PointLomaNU
Record Dates: First submitted 2025-04-26; First posted 2025-06-05 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Injury;Sports; Muscle Soreness
Keywords: kinematics; kinetics; electromyography
MeSH Terms: conditions — Athletic Injuries; Myalgia

STUDY DESIGN:
Intervention Model Description: This cross-sectional trial involves a single visit with two sessions of data collection in which performance of each participant will be assessed before and after a treatment session.
  * Test 1: passive range-of-motion (ROM) and 3D motion capture
  * Intervention: control group (flexibility and stretching treatment); intervention (flexibility and stretching treatment with percussive therapy)
  * Test 2: passive range-of-motion (ROM) and 3D motion capture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No percussive therapy will be applied to participants in this group.
- Intervention (Experimental): Percussive therapy will be applied to participants in this group.
  Interventions: Device: Theragun Prime

INTERVENTIONS:
Device: Theragun Prime — Percussion massager
  Arms: Intervention

SUMMARY:
With increased demand on pickleball as a recreational exercise, it is of interest in investigating the biomechanical characteristics of pickleball and determining the impacts of percussion therapy on them. This study aims to examine the effects of percussion therapy on the biomechanics of pickleball movement and muscle activation patterns in recreational pickleball players. It is hypothesized that kinematics and kinetics of pickleball performance improves after 4 weeks of percussion therapy.

DETAILED DESCRIPTION:
Pickleball has rapidly increasing its playing population among people with different ages and performance levels. While pickleball is keeping people of all age active, injury prevalence of recreational pickleball players particularly for elderly populations has rapidly become a great concern in health care in recent years. It is crucial not only for individuals who play the sports but also for sports medicine professionals to prevent injuries and assure wellbeing of pickleball players. Percussion therapy with a handheld massage gun has widely utilized both in clinical or sports settings and by individuals as a self-care device, allowing the treatment popular and accessible. While previous research has examined acute effects of percussion therapy, the impacts of percussion therapy on exercise performance are not yet fully understood mainly due to diverse designs, protocols, and qualities of previous studies. Moreover, little is known how biomechanical characteristics (i.e., joint kinematics and kinetics) of sports specific movements of pickleball are altered after the percussion therapy. With Increased demand on pickleball as a recreational exercise, it is of interest in investigating the biomechanical characteristics of pickleball and determining the impacts of percussion therapy on them. The proposed project aims to examine the effects of percussion therapy on the biomechanics of pickleball movement and muscle activation patterns in recreational pickleball players. It is hypothesized that kinematics and kinetics of pickleball performance improves as well as static joint range of motion (ROM) after the percussion therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18 - 80 years old
* Free from injury in lower extremity for the last 6 months
* Plays pickleball regularly defined as self-reported participation on at least a weekly basis for a year or more

Exclusion Criteria:

* Joint injury within previous 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Passive hip flexion range-of-motion (ROM) | Cross-sectional design with two tests over a 30 minute period (before and after a 20 minute intervention session)
  Passive flexion ROM (degrees) of the dominant hip
Passive knee flexion range-of-motion (ROM) | Cross-sectional design with two tests over a 30 minute period (before and after a 20 minute intervention session)
  Passive flexion ROM (degrees) of the dominant knee
Peak hip extensor moment | Cross-sectional design with two tests over a 30 minute period (before and after a 20 minute intervention session)
  Peak extensor moment (Nm) of the dominant hip during change-of-direction tasks
Peak hip abductor moment | Cross-sectional design with two tests over a 30 minute period (before and after a 20 minute intervention session)
  Peak abductor moment (Nm) of the dominant hip during change-of-direction tasks
Peak knee extensor moment | Cross-sectional design with two tests over a 30 minute period (before and after a 20 minute intervention session)
  Peak extensor moment (Nm) of the dominant knee during change-of-direction tasks
Peak knee abduction moment | Cross-sectional design with two tests over a 30 minute period (before and after a 20 minute intervention session)
  Peak abduction moment (Nm) of the dominant knee during change-of-direction tasks

SECONDARY OUTCOMES:
Peak quadriceps group activation intensity | Cross-sectional design with two tests over a 30 minute period (before and after a 20 minute intervention session)
  Peak muscle activation via surface electromyography (EMG) as normalized by the maximum voluntary isometric contraction (% MVIC) of the dominant quadriceps (rectus femoris, vastii muscles) during change-of-direction tasks
Peak lateral hamstrings group activation intensity | Cross-sectional design with two tests over a 30 minute period (before and after a 20 minute intervention session)
  Peak muscle activation via surface electromyography (EMG) as normalized by the maximum voluntary isometric contraction (% MVIC) of the dominant lateral hamstrings (biceps femoris, semitendinosus muscles) during change-of-direction tasks

CONTACTS AND LOCATIONS:
Locations (1):
- PLNU x Padres Biomechanics Laboratory, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share the data after study completion.

REFERENCES:
- [Result] Ates R, Yasar P, Baskurt F, Baskurt Z, Ercan S. A Comparison of the Acute Effects of Percussion Massage Therapy and Static Stretching on Hamstring Elasticity. Ethiop J Health Sci. 2023 Jul;33(4):695-702. doi: 10.4314/ejhs.v33i4.16. PMID 38784209
- [Result] Azar FM, Lamplot JD, Bernholt DL, Spence DD. Pickleball: A Standard Review of Injury Prevalence and Prevention in a Rapidly Growing Sport. J Am Acad Orthop Surg. 2024 Nov 15;32(22):e1130-e1141. doi: 10.5435/JAAOS-D-24-00151. Epub 2024 Jul 26. PMID 39079099
- [Result] Alvarado F, Valenzuela KA, Finn A, Avila EL, Crussemeyer JA, Nakajima M. The Biomechanical Effects of Percussive Therapy Treatment on Jump Performance. Int J Exerc Sci. 2022 Jul 1;15(1):994-1006. doi: 10.70252/UIIY1243. eCollection 2022. PMID 36161205
- [Result] Liu Z, Zhong Y, Maemichi T, Zhou Q, Okunuki T, Li Y, Kazuki W, Kumai T. Acute Effects of Local High-Frequency Percussive Massage on Deep Fascial and Muscular Stiffness and Joint Range of Motion in Young Adult Men. J Sport Rehabil. 2024 Mar 20;33(4):252-258. doi: 10.1123/jsr.2022-0455. Print 2024 May 1. PMID 38508160
- [Result] Sams L, Langdown BL, Simons J, Vseteckova J. The Effect Of Percussive Therapy On Musculoskeletal Performance And Experiences Of Pain: A Systematic Literature Review. Int J Sports Phys Ther. 2023 Apr 1;18(2):309-327. doi: 10.26603/001c.73795. eCollection 2023. PMID 37020441